CLINICAL TRIAL: NCT02645422
Title: Genetic Determinants and Clinical Consequences of Early-onset Severe Obesity
Acronym: PeLi
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Folkhälsan Researech Center (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Petra Loid, MD, Helsinki University Central Hospital
Other Study IDs: HUCH43/2015
Record Dates: First submitted 2015-12-09; First posted 2016-01-01 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study is to identify new obesity-related genetic defects and determine their association with clinical manifestations in families with childhood-onset severe obesity. The investigators hypothesize that by exploring children with severe early-onset obesity they can find new obesity-related genetic defects and by exploring obesity-associated clinical manifestations the investigators can elucidate the outcomes of severe childhood obesity.

DETAILED DESCRIPTION:
Obesity is a complex disorder with many contributing genetic and environmental factors. The genetic causes and mechanisms for severe childhood obesity are still incompletely understood. It is acknowledged that obesity in some individuals could be a consequence of rare genetic variants with strong effect - these rare variants might be population specific.

The aims of this study are to determine

* inheritance patterns of early-onset obesity
* new obesity-related genetic variants and disease-causing gene mutations
* the association between obesity-related genetic defects and clinical manifestations
* the association between obesity-related genetic defects and psychiatric symptoms

in patients with early-onset obesity and their first-degree relatives

Significant advancements in genetic methodology provide new tools to explore genetic defects underlying obesity. Family-based approach provides several advantages compared to cohort studies to investigate genetic determinants of complex diseases.The unique genetic composition of the Finnish population enables identification of novel genetic entities.

Discovery of genetic defects associated with severe childhood-onset obesity will increase the investigators understanding of the pathogenesis of obesity and allows early detection, by genetic testing, of those at increased risk and optimal targeting of preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents age 10-18 years
* height-adjusted weight >60 % before the age of 7 years.
* Finnish descent

Exclusion Criteria:

* patients with a known endocrine or genetic disorder underlying obesity (e.g. Prader-Willi syndrome, hypercortisolism, hypothyroidism)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study subjects include children and adolescent with severe, early-onset childhood obesity. Early-onset obesity is defined as height-adjusted weight >60 % (corresponding to severe obesity) before the age of 7 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2023-09-22 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with gene mutations or genetic variants in children with early-onset severe obesity | Baseline, first day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Outi Mäkitie, Prof., Study Director — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No